CLINICAL TRIAL: NCT04117516
Title: Safety and Efficacy of Percutaneous Carpal Tunnel Release Versus Open Surgery: a Randomized Clinical Trial.
Brief Title: Safety and Efficacy of Percutaneous Carpal Tunnel Release Versus Open Surgery
Acronym: CATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Javier Coloma, Principal Investigator, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COTHAV1
Record Dates: First submitted 2019-08-11; First posted 2019-10-07 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Percutaneous carpal tunnel release
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Conversion to Open Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open surgery (Active Comparator): 30 patients will be operated with an open carpal tunnel release.
  Interventions: Procedure: Open surgery
- Percutaneous surgery (Experimental): 30 patients will be operated with a percutaneous carpal tunnel release.
  Interventions: Procedure: Percutaneous surgery

INTERVENTIONS:
Procedure: Open surgery — Open carpal tunnel release will be performed, in the theatre, with tourniquet, under local anesthesia and sedation, through a short longitudinal volar "classical" approach of the hand, that allows to visualize the complete division of the ligament.
  Arms: Open surgery
Procedure: Percutaneous surgery — Percutaneous carpal tunnel release will be performed, ambulatory, with a percutaneous scalpel, through a short transverse volar approach, 1-2cm proximal to the wrist, under Wide Awake Local Anesthesia with No Tourniquet.
  Arms: Percutaneous surgery

SUMMARY:
Hypothesis: Percutaneous ambulatory carpal tunnel release offers similar outcomes to the open approach in the theatre.

Study design: Two-groups randomized single-blind interventional non-inferiority clinical trial.

DETAILED DESCRIPTION:
Background: Carpal tunnel syndrome (CTS) is the most common compressive neuropathy in the upper limb, with a prevalence of around 1'14% and 14'4% of the population.

The clinical symptoms are usually pain, paresthesias and numbness on the sensitive distribution territory of the median nerve in the hand.

Conservative treatment is used for the mild cases, and surgery for the moderate and severe ones, or when the conservative treatment has failed.

Open carpal tunnel release is the gold standard surgery, with a short longitudinal volar approach that allows to visualize the complete division of the ligament.

Over the last few years, endoscopic techniques have been introduced, offering some advantages such as: lower postoperative pain, earlier return to work and less complications due to the wound. Despite this, it has not been popularised, probably, because it is a challenging and more expensive surgical procedure.

Based on the minimally invasive endoscopic approach, and with the aim of obtaining the same benefits, and avoid the complications of the open surgery, several devices have been developed to perform a percutaneous release.

Hypothesis: Percutaneous ambulatory carpal tunnel release offers similar outcomes to the open approach in the theatre.

Study design: Two-groups randomized single-blind interventional non-inferiority clinical trial.

Methods: Sixty patients reporting CTS symptoms, that are confirmed by clinical exam and nerve conduction studies, will be included. Participants will be randomized in two arms. Patients from one group will be operated with an open carpal tunnel release, in the theatre, with tourniquet, under local anesthesia and sedation, through a short longitudinal volar "classical" approach of the hand, that allows to visualize the complete division of the ligament. The other group will be operated with a percutaneous approach, ambulatory, with a short transverse volar approach, 1-2cm proximal to the wrist, under Wide Awake Local Anesthesia with No Tourniquet.

The main outcome measures will be the Boston Carpal Tunnel Questionnaire, Quick DASH questionnaire, Douleur Neuropathique 4 questions, Visual Numeric Scale and grip strength. The scales and questionnaires will be administrated to participants preoperative, 4 weeks and 24 weeks postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old.
* Positive electromyography, confirming carpal tunnel syndrome.
* Capable to understand risks and advantages of both procedures.
* Normal blood tests.

Exclusion Criteria:

* Previous carpal tunnel release in the same hand.
* Previous fracture or dislocation in the area around the forearm, wrist or hand.
* Signs or symptoms of infection.
* Psychiatric disorders.
* Antiplatelet or anticoagulant therapy, that cannot be suspended due to underlying pathology, and does not allow the surgery to be performed.
* Coagulation disorders, or any underlying pathology, with high risk of thrombosis or bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Boston Carpal Tunnel Questionnaire | Preoperative, 4 weeks and 24 weeks after surgery.
  Outcomes from both interventions will be measured with this symptom severity and functional status carpal tunnel specific scale.
  The range of the final results are from 19 (no symptoms) to 95 (severe symptoms).

SECONDARY OUTCOMES:
Visual Numeric Scale | Preoperative, 4 weeks and 24 weeks after surgery.
  Pain relief will be measured with the VNS. The range of the scale is from 0 (no symptoms) to 10 (severe symptoms).
Quick-DASH (Disabilities of Arm, Shoulder and Hand) | Preoperative, 4 weeks and 24 weeks after surgery.
  Disabilities of the hand will be measured with Quick-DASH. The range of the final results are from 0 (no symptoms) to 100 (severe symptoms).
Douleur Neuropathique 4 questions (DN4) | Preoperative, 4 weeks and 24 weeks after surgery.
  Neuropathic pain relief with the DN4. The range of the final results are from 0 (no symptoms) to 10 (severe symptoms).
  A result of more than 4 indicates neuropathic pain.
Consumer Reports Effectiveness Scale (CRES-4) | 24 weeks after surgery.
  Patient´s satisfaction after the procedures The range of the final results are from 0 to 300. A higher score indicates a better outcome of the treatment for the patient.
Time off work | 24 weeks after surgery.
  Differences in time off work between both procedures measured in days.
Grip strength | Preoperative, 4 weeks and 24 weeks after surgery.
  Measured in Kilograms with a "Deyard EH101" dynamometer
Number of other complications | 4 weeks and 24 weeks after surgery.
  Any complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Arnau de Vilanova/Lliria, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided